CLINICAL TRIAL: NCT01970670
Title: Contrast-Enhanced Digital Mammography (CEDM) vs Contrast-Enhanced Breast MRI (CE-MRI) in Patients With Known Breast Cancer
Brief Title: Contrast-Enhanced Digital Mammography(CEDM) vs Contrast-Enhanced Breast MRI(CE-MRI) in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: BRS0031; 27277
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Breast - Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective is to determine how accurately one can estimate the size of the index tumor on preoperative imaging in patients with known breast cancer, using pathology as a reference standard. The primary endpoint, which will be measured on CEDM,and CE-MRI, is the maximum diameter (mm) of the index tumor.

DETAILED DESCRIPTION:
The primary objective is to determine how accurately one can estimate the size of the index tumor on preoperative imaging in patients with known breast cancer, using pathology as a reference standard. The primary endpoint, which will be measured on CEDM,and CE-MRI, is the maximum diameter (mm) of the index tumor.

ELIGIBILITY:
Identify inclusion criteria

1. Histologically confirmed invasive and/or in situ carcinoma of the breast
2. Any race and ethnicity
3. Females 18-70 years of age
4. Willing and able to provide informed consent
5. Subject will have a CE-MRI exam within one month (31 days) of enrolling or has had a CE-MRI exam within one month (31 days) prior to enrolling with no interval treatment or procedure between the CEDM and CE-MRI

Identify exclusion criteria

1. Unwilling or unable to undergo informed consent
2. Planned to undergo neoadjuvant chemotherapy
3. Breast implants
4. Pregnant (NOTE: If subject is unsure of pregnancy status, a pregnancy test will be performed for confirmation.)
5. Breast-feeding
6. Surgical excision of the biopsy proven malignancy
7. Known allergy to gadolinium contrast agents
8. Contraindication for MRI (ex: pacemaker, ferromagnetic aneurysm clips or other ferromagnetic surgical implant or severe claustrophobia)
9. Suspected to be at risk to complications from the contrast agent. These include the standard iodinated contrast agent contraindications:

   1. Subject has renal insufficiency as determined by an elevated serum creatinine and is not being treated with dialysis.
   2. Documentation of a normal eGFR (MDRD) within the previous 2 months will be required for any subject with any of the following risk factors for renal insufficiency:

   i. Age > 70 ii. Diabetes iii. Personal history of renal disease iv. Family history of renal disease (e.g., polycystic kidney disease) v. Known solitary kidney vi. Other medical conditions that may affect the kidney (e.g., Lupus, multiple myeloma) c. Subject has taken metformin (Glucophage) within 48 hours of procedure d. Subject has had a prior reaction to iodinated contrast e. Subject has multiple allergies and/ or severe asthma regularly treated with medication f. Subject has had an episode of serious allergic reaction (anaphylaxis) to any substance

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women, ages18-70 years old, of any race and ethnicity, with a recent diagnosis of breast cancer (histologically confirmed invasive and/or in situ carcinoma of the breast)who have not undergone surgery, are not planned to undergo neoadjuvant chemotherapy; and have a CE-MRI within 1 month(31 days) of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2017-02-17 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Number of partipicants with adverse events | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jafi Lipson, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States